CLINICAL TRIAL: NCT03573388
Title: OMEF: Optical-coherence-tomography (OCT) Measures Predicting Fractional-flow-reserve (FFR)
Brief Title: OCT Measures Predicting FFR
Acronym: OMEF
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Burzotta, MD, PhD, Catholic University of the Sacred Heart
Other Study IDs: 20042018
Record Dates: First submitted 2018-04-23; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Coronary Disease
Keywords: Intermediate coronary lesions; Fractional flow reserve; Optical coherence tomography
MeSH Terms: conditions — Coronary Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Optical coherence tomography (OCT)
  Interventions: Device: Optical coherence tomography (OCT)

INTERVENTIONS:
Device: Optical coherence tomography (OCT) — Lesion OCT assessment

SUMMARY:
Background: the decision-making process of patients with angiographically-intermediate coronary lesions (ICL) is clinically challenging and may benefit from adjunctive invasive techniques. Fractional-flow-reserve (FFR) represents the gold standard to evaluate ICL but optical-coherence-tomography (OCT) is a novel, promising, high resolution coronary imaging technique.

Objectives:

1. Investigate the relation between OCT and FFR parameters in ICL and understand if OCT measures may predict FFR.
2. Understand if OCT parameters may predict clinical outcome of patients with ICL not underwent revascularization on the bases of negative FFR.

Study design: multicentre, international, individual patient's level data pooled analysis.

DETAILED DESCRIPTION:
Principal investigators that enrolled stable or unstable patients with ICL who underwent both FFR and OCT assessment of the same lesion, will be contacted to participate the study. Agreeing investigators will be asked to complete a structured database by providing a series of key baseline clinical and angiographic data, OCT and FFR parameters.

Collected dataset will include: sex, age, hypertension, diabetes, hypercholesterolemia, current smoking, family history of CAD, clinical presentation, previous PCI, previous MI, previous CABG, non-invasive ischemia, angina, n° of diseased vessels, diseased vessel, percentage diameter stenosis at quantitative coronary angiography (QCA% stenosis), length of stenosis at quantitative coronary angiography, presence of thrombus or ulceration, MLA, area stenosis at OCT, FFR protocol (intracoronary adenosine, endovenous adenosine, contrast) results and long term clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angiographically-intermediate coronary lesion
* Patients who underwent both FFR and OCT assessment of the same lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable or unstable patients with intermediate coronary lesions who underwent both FFR and OCT assessment of the same lesion
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
OCT measures predicting FFR - mean lumen area | 1 day
  ICL mean lumen area (MLA)
OCT measure predicting FFR - area stenosis | 1 day
  ICL percentage area stenosis (AS)
OCT measure predicting FFR - thrombus or ulceration | 1 day
  Presence of thrombus or ulceration at the level of ICL

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) in untreated patients (no PCI or CABG) | 1 year
  Major Adverse Cardiac Events (MACE) defined as the composite of:
  * cardiac death (any death not clearly attributed to non cardiac causes)
  * (spontaneous) myocardial infarction (MI)
  * surgical or percutaneous coronary revascularization of the target lesion (PCI o CABG)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico A. Gemelli. Università Cattolica del Sacro Cuore, Roma, Italy

REFERENCES:
- [Derived] Lombardi M, Vergallo R, Costantino A, Bianchini F, Kakuta T, Pawlowski T, Leone AM, Sardella G, Agostoni P, Hill JM, De Maria GL, Banning AP, Roleder T, Belkacemi A, Trani C, Burzotta F. Development of machine learning models for fractional flow reserve prediction in angiographically intermediate coronary lesions. Catheter Cardiovasc Interv. 2024 Sep;104(3):472-482. doi: 10.1002/ccd.31167. Epub 2024 Aug 1. PMID 39091119